CLINICAL TRIAL: NCT07165288
Title: Effect of Continuous Midwifery Support on Comfort, Sleep Quality, and Breastfeeding Self-Efficacy in Primiparous Women: A Follow-Up Study From Pregnancy to Motherhood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palu Devlet Hastanesi (Other)
Responsible Party: Principal Investigator, Sümeyye ŞİMŞEK, Midwife / MSC Student, Palu Devlet Hastanesi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Palu Devlet Hastanesi
Record Dates: First submitted 2025-03-08; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-03

CONDITIONS: Effect of Continuous Midwifery Support on Comfort, Sleep, and Breastfeeding Self-Efficacy in Primiparous Women: A Follow-Up From Pregnancy to Motherhood
Keywords: Breastfeeding self-efficacy; Comfort; Continuous midwifery support; Primiparity; Sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous midwife support care (Active Comparator): Experimental Group First Interview (36th week of pregnancy - first encounter) Second Interview (37th week of pregnancy) Third Interview (38th week of pregnancy) Fourth Observation (Hospital follow-up covering the labor process and the first day after birth)
  Fifth Interview (5-7th day after birth):
  Interventions: Other: Continuous midwife support care; Other: Pilates ball usage; Other: warm shower
- Control Group (No Intervention): Control Group First Interview (36th week of pregnancy - first encounter)
  Second Interview (5-7th day after birth):

INTERVENTIONS:
Other: Continuous midwife support care — Primiparous pregnant women are provided with continuous and individual midwife support starting from the 36th week until the postpartum period.
  Arms: Continuous midwife support care
Other: Pilates ball usage — Primiparous pregnant women were provided with educational support starting from the prenatal period to the postnatal period. In addition, depending on the preferences of the pregnant woman, at least one of the above-mentioned practices was chosen with the accompaniment of a midwife at the time of birth.
  Arms: Continuous midwife support care
Other: warm shower — It was generally applied to the majority of our pregnant women within the scope of training.
  Arms: Continuous midwife support care

SUMMARY:
The study was conducted to determine the effect of continuous midwife support provided to primiparous pregnant women until the postpartum period on comfort, sleep quality and breastfeeding self-sufficiency.

DETAILED DESCRIPTION:
The study was conducted to determine the effect of continuous midwifery support provided to primiparous pregnant women until the postpartum period on comfort, sleep quality, and breastfeeding self-efficacy.

Materials and Methods: This randomized controlled trial included a total of 128 pregnant women-64 in the experimental group and 64 in the control group-who were in the 36th week of pregnancy and applied to the Elazığ Palu State Hospital Gynecology and Obstetrics Outpatient Clinic. During the first interview (36th week), pre-test data were collected in the NST room using the "Personal Information Form", "General Comfort Questionnaire", "Pittsburgh Sleep Quality Index", and the "Antenatal Breastfeeding Self-Efficacy Scale-Short Form".

In the second (37th week of pregnancy), third (38th week of pregnancy), and fifth interviews (within the first 4-8 hours postpartum), participants in the experimental group received training in line with educational booklets prepared by the researcher. Since the fourth interview was scheduled during the labor process, continuous support was provided to the pregnant women during childbirth. The sixth interview was conducted between the 5th and 7th days postpartum, during which post-test data were collected using the "General Comfort Questionnaire", "Pittsburgh Sleep Quality Index", and the "Postnatal Breastfeeding Self-Efficacy Scale-Short Form".

ELIGIBILITY:
Inclusion Criteria:

All pregnant women who communicate verbally and do not have a reading or writing disability,

* Having a singleton healthy pregnancy,
* Having a primiparous pregnancy in the 36th week of pregnancy,
* Not a midwife by profession,
* Not having any diagnosed psychiatric problems were included.

Exclusion Criteria:

* Women who developed an indication for cesarean section were excluded.

For postpartum women;

* Those who developed a condition requiring separation from their babies,
* Those who wanted to leave the study during the follow-ups,
* Those who filled out the data collection forms incompletely,
* Those who gave birth before the third interview were excluded.

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Since the study will be conducted with pregnant women, only female individuals are eligible to participate.
Enrollment: 128 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
It was determined that continuous midwife support provided to primiparous pregnant women until the postpartum period increased women's comfort, sleep quality and breastfeeding self-sufficiency. | 8 weeks
  Outcome Measure Title:
  General Comfort Level
  Description:
  General comfort level is assessed using the General Comfort Scale developed by Kolcaba (1992) and validated in Turkish by Kuğuoğlu and Karabacak (2008). This 48-item Likert-type scale includes four subdimensions: Physical Comfort (12 items), Psychospiritual Comfort (13 items), Environmental Comfort (13 items), and Sociocultural Comfort (10 items). Scores are calculated by reverse coding negative items, summing with positive items, and dividing by the number of items to yield an average score ranging from 1 (low comfort) to 4 (high comfort). Reliability coefficients (Cronbach's alpha) in this study were 0.773 (experimental group) and 0.905 (control group).
  Measurement Unit:
  Mean score (1-4),
It was determined that continuous midwife support provided to primiparous pregnant women until the postpartum period increased women's comfort, sleep quality and breastfeeding self-sufficiency. | 8 weeks
  Title: Sleep Quality Measured by the Pittsburgh Sleep Quality Index (PSQI) Description: Sleep quality was assessed using the PSQI, a validated questionnaire measuring sleep quality over the past month. The scale consists of 19 self-reported items scored from 0 to 3, with total scores ranging from 0 to 21. Scores above 5 indicate poor sleep quality. The study measured the change in PSQI total scores from baseline (pre-intervention) to post-intervention between the experimental and control groups.
It was determined that continuous midwife support provided to primiparous pregnant women until the postpartum period increased women's comfort, sleep quality and breastfeeding self-sufficiency. | 8 weeks
  Title: Breastfeeding Self-Efficacy Measured by the Antenatal Breastfeeding Self-Efficacy Scale - Short Form (AEBS-SF) Description: Breastfeeding self-efficacy was evaluated using the AEBS-SF, a validated 14-item questionnaire with a 5-point Likert scale (1 = Not confident at all, 5 = Always confident). Scores range from 14 to 70, with higher scores indicating greater breastfeeding self-efficacy. The study assessed changes in breastfeeding self-efficacy scores from baseline to post-intervention in the experimental group.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyye ŞİMŞEK, MSC student, Principal Investigator — İnönü Üniversitesi
Locations (1):
- Palu Devlet Hastanesi, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I think this is a special work. So I am undecided about it.

REFERENCES:
- See also: Qualitative study in a maternity unit in Norway, where approximately 4000 births take place each year. In-depth interviews were conducted with ten midwives working in two different maternity units. Qualitative data were analysed using systematic text con — https://pubmed.ncbi.nlm.nih.gov/26370160/
- Available data/document: Study Protocol: different example — https://pubmed.ncbi.nlm.nih.gov/23473911/ — Our study found that the support provided had a significant impact on primiparous mothers.